CLINICAL TRIAL: NCT00271765
Title: A Phase II Randomized, Placebo-Controlled, Single-Blind, Multi-Center Dose-Escalation Study to Evaluate Tolerability, Safety, Pharmacokinetics, and Pharmacodynamics of a Single Intravenous Administration of INO-1001 in Subjects With ST-Elevation Myocardial Infarction Undergoing Primary Percutaneous Coronary Intervention
Brief Title: A Study of INO-1001, an Intravenous PARP (Poly [ADP Ribose] Polymerase) Inhibitor in Acute Heart Attack Patients Undergoing Primary Percutaneous Coronary Intervention
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Inotek Pharmaceuticals Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IPC-15-2003
Record Dates: First submitted 2006-01-03; First posted 2006-01-04 (Estimated); Last update posted 2006-11-29 (Estimated); Status verified 2006-11

CONDITIONS: Acute Myocardial Infarction
Keywords: Myocardial infarction; Coronary angioplasty; PARP inhibitor; PARP inhibition; Heart Attack
MeSH Terms: conditions — Myocardial Infarction | interventions — INO 1001

INTERVENTIONS:
Drug: INO-1001

SUMMARY:
The primary purpose of this study is to assess the safety of INO-1001 in subjects who have experienced a heart attack and are to be treated with coronary angioplasty.

DETAILED DESCRIPTION:
Currently, heart attacks may be treated with clot-dissolving medicines, coronary angioplasty, or a combination of both. Unblocking of blood flow to the heart following coronary angioplasty can cause side effects such as heart tissue and blood vessel damage, abnormal heart rhythms and death of heart muscle cells.

In animal studies, the PARP enzyme has been shown to be involved in damaging heart muscle after the sudden unblocking of coronary arteries. INO-1001 blocks the PARP enzyme, and so it may reduce heart damage in humans who have had their coronary arteries unblocked after a heart attack.

A total of 40 patients will be selected and randomly assigned to either INO-1001 or placebo (sugar water). One dose only of the drug will be given prior to coronary angioplasty. Patients will be followed until 30 days after surgery.

The following information will be gathered: vital signs, symptoms, physical examination, blood and urine tests, electrocardiograms, and other information from medical charts.

The information provided in this listing is disclosed solely to comply with regulatory requirements. The drug INO-1001 has not yet been approved for marketing and is only available to patients who participate in a clinical trial and are chosen for the treatment group.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with acute myocardial infarction (as defined in protocol) with onset within 24 hours prior to randomization.
* Scheduled for primary percutaneous coronary intervention within 3 hours of presentation at a hospital participating in this study.
* Males and non-pregnant, non-lactating females.

Exclusion Criteria:

* Subjects will be required to undergo a full medical review in order to exclude serious medical, or psychological illness prior to inclusion.
* History of a hypersensitivity reaction to more than three drugs or mannitol.
* Participation in any investigational study within 30 days of randomization
* Treatment with certain restricted medications within a specified time prior to participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2004-01; Study Completion 2006-06

PRIMARY OUTCOMES:
The safety of INO-1001 will be measured by evaluation of symptoms, vital signs, physical examination, laboratory data, electrocardiograms, etc.

SECONDARY OUTCOMES:
The effect of INO-1001 on heart muscle damage will be evaluated by blood tests. Other blood tests will measure how INO-1001 is absorbed and removed by the body after exposure to different doses.

CONTACTS AND LOCATIONS:
Locations (16):
- United States (10):
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Porter Hospital, Valparaiso, Indiana
  - St. Paul Heart Clinic, Saint Paul, Minnesota
  - Newark, New Jersey
  - Toledo Hospital, Toledo, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Black Hills Cardiovascular Research, Rapid City, South Dakota
  - Burlington, Vermont
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - West Virginia University, Morgantown, West Virginia
- Israel (6):
  - Rambam Medical Center, Haifa
  - Meir Medical Center, Kfar Saba
  - Hasharon Medical Center, Petah Tikva
  - Rabin Medical Center, Petah Tikva
  - Rehovot
  - Assaf Harofe Medical Centre, Ẕerifin

REFERENCES:
- [Background] Liaudet L, Szabo E, Timashpolsky L, Virag L, Cziraki A, Szabo C. Suppression of poly (ADP-ribose) polymerase activation by 3-aminobenzamide in a rat model of myocardial infarction: long-term morphological and functional consequences. Br J Pharmacol. 2001 Aug;133(8):1424-30. doi: 10.1038/sj.bjp.0704185. PMID 11498530
- [Background] Zingarelli B, Cuzzocrea S, Zsengeller Z, Salzman AL, Szabo C. Protection against myocardial ischemia and reperfusion injury by 3-aminobenzamide, an inhibitor of poly (ADP-ribose) synthetase. Cardiovasc Res. 1997 Nov;36(2):205-15. doi: 10.1016/s0008-6363(97)00137-5. PMID 9463632
- [Background] Zingarelli B, Salzman AL, Szabo C. Genetic disruption of poly (ADP-ribose) synthetase inhibits the expression of P-selectin and intercellular adhesion molecule-1 in myocardial ischemia/reperfusion injury. Circ Res. 1998 Jul 13;83(1):85-94. doi: 10.1161/01.res.83.1.85. PMID 9670921
- [Background] Grupp IL, Jackson TM, Hake P, Grupp G, Szabo C. Protection against hypoxia-reoxygenation in the absence of poly (ADP-ribose) synthetase in isolated working hearts. J Mol Cell Cardiol. 1999 Jan;31(1):297-303. doi: 10.1006/jmcc.1998.0864. PMID 10072736
- [Derived] Morrow DA, Brickman CM, Murphy SA, Baran K, Krakover R, Dauerman H, Kumar S, Slomowitz N, Grip L, McCabe CH, Salzman AL. A randomized, placebo-controlled trial to evaluate the tolerability, safety, pharmacokinetics, and pharmacodynamics of a potent inhibitor of poly(ADP-ribose) polymerase (INO-1001) in patients with ST-elevation myocardial infarction undergoing primary percutaneous coronary intervention: results of the TIMI 37 trial. J Thromb Thrombolysis. 2009 May;27(4):359-64. doi: 10.1007/s11239-008-0230-1. Epub 2008 Jun 6. PMID 18535785